CLINICAL TRIAL: NCT04867291
Title: Seaweed, the Food Matrix, and Iodine Bioavailability
Acronym: IoBio
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Glasgow (Other)
Responsible Party: Principal Investigator, Emilie Combet, Senior Lecturer in Nutrition, University of Glasgow
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 200180075
Record Dates: First submitted 2021-04-27; First posted 2021-04-30 (Actual); Last update posted 2021-04-30 (Actual); Status verified 2021-04

CONDITIONS: Iodine Bioavailability
MeSH Terms: interventions — PIZZA protein, Arabidopsis; Potassium Iodide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Pizza (Experimental): Consumption of a portion of Eat Balanced pizza equivalent to 200 µg of iodine (half a pizza) consumed with 450 mL water. Collection of urine for 36 hours following pizza ingestion. Collection of one fecal sample up to 24 hours following pizza ingestion.
  Interventions: Dietary Supplement: Pizza
- Seaweed Sheets (Experimental): Consumption of a portion of Itsu Crispy Seaweed Thins equivalent to 200 µg of iodine (10g) consumed with 450 mL water. Collection of urine for 36 hours following ingestion. Collection of one fecal sample up to 24 hours following ingestion.
  Interventions: Dietary Supplement: Seaweed Sheets
- Seaweed Powder (Experimental): Consumption of a portion of seaweed powder in a capsule equivalent to 200 µg of iodine (0.25g) consumed with 450 mL water. Collection of urine for 36 hours following ingestion. Collection of one fecal sample up to 24 hours following ingestion.
  Interventions: Dietary Supplement: Seaweed Powder
- Potassium Iodide Supplement (Experimental): Consumption of a portion of Piping Rock Potassium Iodide supplements equivalent to 200 µg of iodine (1.3 tablets) consumed with 450 mL water. Collection of urine for 36 hours following ingestion. Collection of one fecal sample up to 24 hours following ingestion.
  Interventions: Dietary Supplement: Potassium iodide

INTERVENTIONS:
Dietary Supplement: Pizza — Portion equivalent to 200 µg of iodine (half a pizza), consumed with ~450mL of water.
  Arms: Pizza
Dietary Supplement: Seaweed Sheets — Portion equivalent to 200 µg of iodine (~10g), consumed with two slices of white bread and ~450mL of water.
  Arms: Seaweed Sheets
Dietary Supplement: Seaweed Powder — Portion equivalent to 200 µg of iodine (1 capsule), consumed with two slices of white bread and ~450mL of water.
  Arms: Seaweed Powder
Dietary Supplement: Potassium iodide — Portion equivalent to 200 µg of iodine (1.3 tablets), consumed with two slices of white bread and ~450mL of water.
  Arms: Potassium Iodide Supplement

SUMMARY:
This study explores the influence of the food matrix of seaweed-containing food products on iodine bioavailability. The investigation will ascertain whether iodine bioavailability (as a percentage of the dose ingested that is excreted in urine) is comparable between seaweed sheets, seaweed powder (in capsules), pizza fortified with powdered seaweed, and potassium iodide supplements.

DETAILED DESCRIPTION:
Iodine deficiency can have serious consequences, especially during pregnancy and lactation where the fetus is entirely dependent on its mother for the provision of iodine. There is no current iodine fortification programme in the United Kingdom, and the main sources of iodine are from dietary sources, such as dairy products and seafood. However, seaweed is also a rich source of iodine; the inclusion of iodine (via powdered seaweed) in commonly consumed foods is of potential benefit as a strategy, as it removes the need for consumers to alter their dietary behaviours, which are often culturally standardized.

Seaweed intake (via supplements) can increase the iodine status of women with habitually low-iodine diets. However, reduced bioavailability of iodine from the seaweed matrix has also been displayed, which could impact iodine intake should individuals choose to use seaweed as a dietary source of iodine.

This study tests the influence of the food matrix of seaweed-containing products on iodine bioavailability. This will be evaluated over the course of 27 days, in a randomized crossover trial design with 4 arms. Each arm will be separated by 7 washout days, and participants will follow a low iodine diet (avoiding all seafood, seaweed products, eggs, dairy, fortified plant milk and goitrogens (cabbage, soy etc.) for the 2 days preceding and the 1 day following each feed.

1. Food arm: portion equivalent to 200µg of iodine, half a pizza (Eat Balanced pizza) (consumed with ~450mL of water)
2. Seaweed sheet arm: portion equivalent to 200µg of iodine, ~10g of seaweed sheets (consumed alongside 2 slices of white bread and ~450mL of water)
3. Seaweed powder arm: portion equivalent to 200µg of iodine, 1 capsule (consumed alongside 2 slices of white bread and ~450mL of water).
4. Potassium iodide supplement arm: portion equivalent to 200µg of iodine with ~450mL of water (Piping Rock Potassium Iodide Supplement, consumed alongside 2 slices of white bread)

Iodine excretion will be monitored in urine collected during the 12 hours preceding and 36 hours following the meal. Urine will be collected in 8 timed fractions (0-1h, 1-2h, 2-3h, 3-5h, 5-8h, 8-12h, 12-24h, 24-36h) and participants will be provided with containers and instructions on how to collect their urine. A single fecal sample will also be collected before the first feed, and within 24 hours of all feeds. Participants will also keep a detailed food diary on all study days to enable iodine ingestion monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Premenopausal women
* 18-48 years old
* Signed informed consent

Exclusion Criteria:

* Pregnancy and lactation
* Past and present thyroid conditions/dysfunction
* Allergy to gluten, wheat, or dairy
* Iodine supplement consumption
* Currently taking medication (other than contraceptive)
* Diseases of the gastrointestinal tract
* Current smoker
* Current vegan (pizza contains dairy cheese)
* Having a habitual diet very low in iodine (<1 portion of dairy per day, or <1 portion of fish per week)
* Having a habitual diet very high in iodine (>4 portions of dairy per day, or >4 portions of fish per week)

Ages: 18 Years to 48 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2021-04 (Estimated); Primary Completion 2021-11 (Estimated); Study Completion 2021-11 (Estimated)

PRIMARY OUTCOMES:
Urinary Iodine Excretion (micrograms/L) | 36 hours
  The percentage of iodine ingested from the test foods that is excreted in the 36 hours following test food ingestion will be measured in urine collected fractions: 1-2, 2-3, 3-5, 5-7, 7-12, 12-24, 24-36 hours

SECONDARY OUTCOMES:
Fecal Iodine Excretion (micrograms/g feces) | 24 hours
  The percentage of iodine ingested from the test foods that is excreted in a single fecal sample passed in the 24 hours following test food ingestion

OTHER OUTCOMES:
Gut Bacterial Diversity | Prior to commencement of trial
  Assessed via single fecal sample
Seaweed Fermentation Capacity | Prior to commencement of trial
  Assessment of the capacity of participants' gut microflora to ferment seaweed polysaccharides and release iodine from the food matrix. Assessed via single fecal sample used in an in vitro fermentation model.

CONTACTS AND LOCATIONS:
Overall Officials: Emilie Combet, PhD, Principal Investigator — University of Glasgow

IPD SHARING:
Plan to Share IPD: Undecided